CLINICAL TRIAL: NCT03450278
Title: Effect of Micro-osteoperforation on the Rate of Canine Retraction: A Split Mouth Randomized Controlled Trial
Brief Title: Effect of Micro-osteoperforation on the Rate of Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Aboalnaga, Assistant Lecturer, Dr. Amira Ahmed Mohamed Anis Aboalnaga, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2015-07-10
Record Dates: First submitted 2018-02-13; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Orthodontics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): canine retraction without any means of acceleration.
- micro-osteoperforation (Experimental): canine retraction accelerated with micro-osteoperforation
  Interventions: Procedure: micro-osteoperforation

INTERVENTIONS:
Procedure: micro-osteoperforation — Minor surgical procedure including performance of limited and shallow perforations of the cortical plate of bone to increase the expression of inflammatory cytokines, hence accelerating orthodontic tooth movement.
  Other Names: alveolocentesis; bone puncturing; flapless corticotomy
  Arms: micro-osteoperforation

SUMMARY:
The current study Is a split-mouth Randomized Controlled Trial that was performed to investigate three dimensionally, using digital models and Cone Beam Computed Tomography imaging, the effect of micro-osteoperforations (MOPs) on the rate of tooth movement in a canine retraction model.

DETAILED DESCRIPTION:
Sample size calculation was carried out and resulted in enrolment of 18 female patients requiring bilateral upper first premolars extraction and canine retraction with maximum anchorage. The sample was recruited from the outpatient clinic of the Orthodontic Department, Faculty of Dentistry, Cairo University.

After placement of the fixed orthodontic appliance, leveling and alignment proceeded till 0.016" × 0.022" NiTi upper archwire. Indirect skeletal anchorage was then prepared using TADs inserted bilaterally between the upper 1st molar and 2nd premolar, and the patient was referred for upper 1st premolars extraction.

Three months after extraction, 0.017" × 0.025" stainless-steel upper archwire was inserted and three vertically aligned MOPs were randomly allocated and performed in one side using a single TAD, while the other side served as control. The three MOPs were performed distal to the canine, equidistant in the extraction space. Bilateral canine retraction was then commenced using NiTi closing coil springs delivering 150 gms of force. Before leaving the clinic, a pain questionnaire was given to each patient.

Data were collected from monthly upper impressions, which were poured into stone models and scanned to obtain sequential digital models (T0, T1, T2, T3 & T4), in addition to pre- and post-retraction maxillary CBCT images.

The assessed outcomes were the rate of canine retraction per month, the total distance travelled by the upper canines, first molars anchorage loss, tipping, torque and rotation of upper canines and first molars, canine root resorption and finally the pain related to MOP procedure. Statistical analysis was performed on the gathered data and results were withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* Malocclusion that requires bilateral extraction of the maxillary first premolars and canine retraction with maximum anchorage; Class II division 1 and bimaxillary dentoalveolar protrusion cases.
* Full permanent dentition with exception of the third molars.
* Good oral hygiene and periodontal condition.

Exclusion Criteria:

* Medically compromised patients.
* Patients suffering from any congenital, hereditary or systemic diseases.
* Chronic use of any medications affecting orthodontic tooth movement (e.g. corticosteroids, hormonal therapy, NSAIDs)
* Patients with dental anomalies (e.g. enamel hypoplasia, root dilacerations in maxillary canines).
* Patients with medical conditions that contraindicate surgeries (e.g. bleeding tendency and immunocompromised patients).
* Radiographic evidence of bone loss.

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Rate of maxillary canine retraction | 4 months of canine retraction
  distance (mm) moved by the canine distally per month

SECONDARY OUTCOMES:
Maxillary first molar anchorage loss | 4 months of canine retraction
  anchorage loss (mesial movement) of the maxillary first molar occuring after 4 months of canine retraction.
Maxillary canine tipping, torque and rotation | 4 months of canine retraction
  change in the three dimensional axial inclination (tipping, torque and rotation) of the maxillary canine after 4 months of retraction
Maxillary first molar tipping, torque and rotation | 4 months of canine retraction
  change in the three-dimensional axial inclination (tipping, torque and rotation) of the maxillary first molar after 4 months of canine retraction.
Maxillary canine root resorption | 4 months of canine retraction
  amount of canine root resorption occurred after 4 moths of retraction
Pain caused by the micro-osteoperforation procedure | 1 week after the micro-osteoperforation procedure
  Pain assessed using the Numeric Pain Rating Scale (0-10) assessed immediately after the micro-osteoperforation (MOP) procedure, 1 day, 3 days and 1 week after the MOP procedure. 0 pain score: no pain, (1-3) pain score: mild pain, (3-6) pain scores: moderate pain, (7-10) pain score: severe pain.